CLINICAL TRIAL: NCT06897293
Title: Comparison of Modified Broström Repair + Suture Tape and Modified Broström Repair for CLAI in Chronic Lateral Ankle Instability in Generalized Joint Laxity Cases: A Prospective Cohort Study
Brief Title: Comparison of MBR + Suture Tape and MBR for CLAI in GJL Cases: A Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jiang Dong, Chief physician, Peking University Third Hospital
Other Study IDs: M2024292
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Ankle Sprain; Hypermobility, Joint
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open Modified Broström +Suture tape augmentation group: Patients who accept a modified Broström procedure + Suture tape augmentation operation
  Interventions: Procedure: Modified Broström procedure + Suture tape augmentation operation
- Open Modified Broström group: Patients who accept a modified Broström procedure operation
  Interventions: Procedure: Modified Broström procedure operation

INTERVENTIONS:
Procedure: Modified Broström procedure + Suture tape augmentation operation — Patients with CLAI and GJL will accept the Modified Broström + Suture tape augmentation operation
  Groups: Open Modified Broström +Suture tape augmentation group
Procedure: Modified Broström procedure operation — Patients with CLAI and GJL will accept the Modified Broström procedure operation
  Groups: Open Modified Broström group

SUMMARY:
GJL is a risk factor for postoperative recurrent instability following an MBR for CLAI. Additional suture tape augmentation has been suggested to provide more strength and stability. However, the outcomes of the MBP with suture tape augmentation were unknown, which requires further exploration.

DETAILED DESCRIPTION:
Generalized joint laxity (GJL) is a risk factor for postoperative recurrent instability following an open modified Broström repair (MBR) for chronic lateral ankle instability (CLAI). MBR with suture tape augmentation may provide more strength and stability. However, BPR with suture tape augmentation may lead to rejection of the suture tape. In addition, the outcomes of the MBP with suture tape augmentation were unknown.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lateral ankle instability
* Beighton score ≥4
* Age with 18 to 60 years

Exclusion Criteria:

* Patients with an acute or subacute ankle injury
* Injury of the deltoid ligament
* Alignment of lower extremity greater than 5 degrees
* Fractures of the lower extremity
* Stage III or IV osteoarthritis
* Patients who refused to participate in the study

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients who go to visit a doctor for persistent lateral ankle pain and instability over three months and invalid conservative treatment, with the age of 15 - 55 years. If the Beighton score of the patient is ≥4 and the exclusion criteria are met, he or she is going to be advised to participate in this study.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The American Orthopaedic Foot and Ankle Society (AOFAS) score | postoperative AOFAS score at 1 year
  This score is a primary scale for lateral ankle instability, ranges from 0-100, and the higher of the score is associate with a better outcome.
The American Orthopaedic Foot and Ankle Society (AOFAS) score | postoperative AOFAS score at 2 years
  This score is a primary scale for lateral ankle instability, ranges from 0-100, and the higher of the score is associate with a better outcome.
The American Orthopaedic Foot and Ankle Society (AOFAS) score | postoperative AOFAS score at 6 months
  This score is a primary scale for lateral ankle instability, ranges from 0-100, and the higher of the score is associate with a better outcome.
The American Orthopaedic Foot and Ankle Society (AOFAS) score | postoperative AOFAS score at 3 months
  This score is a primary scale for lateral ankle instability, ranges from 0-100, and the higher of the score is associate with a better outcome.

SECONDARY OUTCOMES:
Anterior displacement and talar tilt angle in stress radiography | postoperative radiographic measures at 2 years
  The outcomes are common indicators for evaluation the lateral stability of ankle, and can be evaluated through same stress radiography
Rate of re-injury | the rate of re-injury at 2 years
  The rate of patients re-sprain after the surgery

OTHER OUTCOMES:
Signal to noise value of anterior talofibular ligament | 6 months post-treatment
  Signal to noise value of the anterior talofibular ligament
Signal to noise value of the anterior talofibular ligament | 12 months post-treatment
  Signal to noise value of the anterior talofibular ligament
Signal to noise value of the anterior talofubular ligament | 24 months post-treatment
  Signal to noise value of the anterior talofibular ligament

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The demographics data, Beighton score, primary and secondary outcomes would be available to other researchers

REFERENCES:
- [Background] Wittig U, Hohenberger G, Ornig M, Schuh R, Reinbacher P, Leithner A, Holweg P. Improved Outcome and Earlier Return to Activity After Suture Tape Augmentation Versus Brostrom Repair for Chronic Lateral Ankle Instability? A Systematic Review. Arthroscopy. 2022 Feb;38(2):597-608. doi: 10.1016/j.arthro.2021.06.028. Epub 2021 Jul 9. PMID 34252562
- [Background] Xu HX, Lee KB. Modified Brostrom Procedure for Chronic Lateral Ankle Instability in Patients With Generalized Joint Laxity. Am J Sports Med. 2016 Dec;44(12):3152-3157. doi: 10.1177/0363546516657816. Epub 2016 Aug 5. PMID 27496909